CLINICAL TRIAL: NCT01676493
Title: A Multicenter, Open-Label, Safety and Pharmacokinetic Study of Oral Codeine Sulfate Administration in Pediatric Subjects 2 Years Old Through 17 Years Old With Post-procedural Pain
Brief Title: A Study of Oral Codeine Sulfate in Pediatric Patients With Post-procedural Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision to stop study due to low recruitment.
Sponsor: Roxane Laboratories (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CODE-OS+T-(2-17)-SPK-1
Record Dates: First submitted 2012-08-24; First posted 2012-08-31 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Codeine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Codeine (Experimental): Codeine Sulfate Oral Solution and Tablet
  Interventions: Drug: Codeine

INTERVENTIONS:
Drug: Codeine
  Other Names: Codeine Sulfate Oral Solution and Tablets

SUMMARY:
This is a multicenter, open-label study to evaluate the safety and PK of oral codeine sulfate in pediatric subjects with mild to moderate post-procedural pain.

DETAILED DESCRIPTION:
Eligible pediatric subjects will complete all screening procedures within 14 days before the scheduled procedure. Screening will be permitted on the day of the procedure. At screening, the subject's parent or guardian will provide written parental permission/informed consent to participate in the study and subjects will provide assent (if required by the local Institutional Review Board [IRB]) before any protocol-specified procedures or assessments are performed.

Subjects may be inpatients, outpatients, or day-surgery patients at the study site who will undergo procedures expected to result in at least mild to moderate post-procedure pain with the day of the procedure noted as Day 0, and will be followed until discharge from the study site.

ELIGIBILITY:
Inclusion Criteria:

1. Has a parent or guardian providing written parental permission/informed consent, with subject assent (if required by local IRB).
2. Is a child 2 years old through 17 years old, inclusive (at the time of informed consent signing).
3. Has a routine pediatric procedure that is expected to cause at least mild to moderate pain.
4. Is expected by the investigator to require a minimum of one (1) dose of oral codeine for the treatment of mild to moderate post-procedural pain.
5. Has the ability to read and understand the study procedures and has the ability to communicate meaningfully with the study investigator and staff (if the subject is of preverbal age or cannot read or communicate meaningfully, then the subject's parent or guardian must meet this criterion).
6. If female subject is of childbearing potential, she must have a negative urine or serum pregnancy test result on the day of the scheduled procedure prior to the procedure. In this population, female of childbearing potential is defined by the onset of menarche, that is, menstruation, whether at irregular or regular intervals (periods).
7. Must have vascular access to facilitate multiple blood draws.

Exclusion Criteria:

1. Is currently lactating.
2. Has significant medical disease(s), laboratory abnormalities, or conditions(s) that in the investigator's judgment could compromise the subject's welfare, ability to communicate with study staff, complete study activities, or would otherwise contraindicate study participation.
3. Weighs less than 10.5 kg. (see Table 4 Maximum Number of Doses of Study Drug by Weight for details)
4. Has weight ≤ 5th or ≥ 95th percentile for age based on CDC Growth Charts. (see Appendix 6)
5. Has received codeine, hydrocodone, morphine or oxycodone in any form in the previous seven (7) days.
6. Has used opioids chronically (e.g., codeine, morphine, oxycodone, hydrocodone, or hydromorphone) for >7 calendar days within the previous 30 days before surgery.
7. Has known hypersensitivity or contraindication to receiving oral opioid(s).
8. Has an active enteral malabsorption disorder.
9. Has impaired liver function (e.g., alanine aminotransferase [ALT] ≥3 times the upper limit of normal [ULN], or bilirubin ≥3 times ULN), known active hepatic disease (e.g., hepatitis), evidence of clinically significant chronic liver disease or other conditions affecting the liver (e.g., chronic hepatitis) that may suggest the potential for an increased susceptibility to hepatic toxicity with oral codeine exposure. NOTE: Subjects with no previous history of liver function impairment may be enrolled before results are available from screening laboratory samples.
10. Has significantly impaired renal function or disease, as evidenced by an estimated glomerular filtration rate (i.e., from creatinine levels using the Schwartz formula) calculated to be less than one-third (1/3) of normal for the applicable age of this study population. NOTE: Subjects with no previous history of kidney function impairment may be enrolled before results are available from screening laboratory samples.
11. Is undergoing a procedure as treatment for acute burns.
12. Has a history of substance abuse or there is evidence of current substance abuse, in the investigator's opinion.
13. Has participated in an interventional clinical study (investigational or marketed product) within 30 days before screening, or plans to participate in another clinical trial in the next 30 days.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
tolerability and safety | up to 24 hours
  * Percentage of subjects who experience any AEs with a causal relationship to the study medication characterized as possible, probable or unknown (unable to judge).
  * Percentage of subjects with SAEs.
  * Percentage of subjects with a UMSS sedation score of 4.
analyte concentrations from blood samples | 24 hours
  Initial Dose of Study Drug
  * Immediately (up to 30 minutes) prior to the dose of oral codeine sulfate.
  * 1 hour (45 to 75 minutes) after administration of the initial dose of oral codeine sulfate.
  * 2 hours (105 to 135 minutes) after administration of the initial dose of oral codeine sulfate.
  Subsequent Doses
  * Immediately (up to 30 minutes) prior to the dose of oral codeine sulfate.
  * 1 hour (45 to 75 minutes) after administration of the dose of oral codeine sulfate.

CONTACTS AND LOCATIONS:
Overall Officials: Dante Landucci, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Children's Medical Center Dallas, Dallas, Texas, United States